CLINICAL TRIAL: NCT02496117
Title: Feasibility of Electrical Mapping and Stimulation of Renal Arteries in Patients Undergoing Renal Denervation
Brief Title: Renal Nerves Stimulation Study
Acronym: RNS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Diagram B.V. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9209
Record Dates: First submitted 2015-07-07; First posted 2015-07-14 (Estimated); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Hypertension; Renal Denervation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: RNS checked RDN
Masking Description: RNS guided RDN
Oversight: Data Monitoring Committee: No

ARMS (2):
- RNS-checked RDN (Active Comparator): 20 patients with hypertension will be enrolled undergoing RNS-checked RDN
  Interventions: Procedure: Electrical mapping, nerve stimulation checked renal denervation procedure
- RNS-guided RDN (Experimental): 20 patients with hypertension will be enrolled undergoing RNS-guided RDN
  Interventions: Procedure: Electrial mapping, nerve stimulation guided renal denervation procedure

INTERVENTIONS:
Procedure: Electrical mapping, nerve stimulation checked renal denervation procedure
  Other Names: RNS-checked RDN
  Arms: RNS-checked RDN
Procedure: Electrial mapping, nerve stimulation guided renal denervation procedure
  Other Names: RNS-guided RDN
  Arms: RNS-guided RDN

SUMMARY:
Study design: Investigator initiated, single centre, feasibility study

Main objectives are twofold:

1. To investigate the feasibility of RNS in patients with therapy resistant hypertension, which is assessing the functional distribution of renal nerves using 3D imaging and differential pacing modalities.
2. To investigate the blood pressure responses and cardiac excitable properties to RNS, and subsequently perform a RDN procedure, guided by 3D mapping by two different techniques e.g. RNS-checked RDN and RNS-guided RDN procedures.

Study population: 40 patients (18 - 80 yr old)

DETAILED DESCRIPTION:
Background: Approximately 10-15% of adults with hypertension are considered to be treatment resistant because their hypertension is uncontrolled despite taking three or more drugs that includes a diuretic. Renal denervation (RDN) is a novel treatment option for therapy resistant hypertension and its rationale originates in denervating the renal sympathetic efferent and afferent coupling with the central autonomic nervous system. By denervating the renal arteries, general sympathetic tone is reduced. Currently, RDN is performed by placing in a spiral pattern 5-6 ablation lesions in each renal artery. 15-30% of the patients do not have any benefit from this procedure. The reason for this is unknown. Experimental data show that renal nerve stimulation (RNS) may serve as a functional endpoint to assess completeness of the RDN procedure. A RNS-guided RDN may prove to be superior to standard RDN (RNS-checked) in blood pressure control.

Main objectives are twofold:

1. To investigate the feasibility of RNS in patients with therapy resistant hypertension, which is assessing the functional distribution of renal nerves using 3D imaging and differential pacing modalities.
2. To investigate the blood pressure responses and cardiac excitable properties to RNS, and subsequently perform a RDN procedure, guided by 3D mapping by two different techniques e.g. RNS-checked RDN and RNS-guided RDN procedures.

Secondary objective:

The secondary objective is to compare both techniques (RNS-checked vs. RNS-guided) in terms of efficacy and safety.

Hypotheses:

* We hypothesize that identification and localization of the sympathetic nerve bundles using 3D navigation systems and selective pacing manoeuvres will allow a functional approach to denervate the kidneys and improve the success rate of this procedure in patients with hypertension.
* We hypothesize that the RNS-guided RDN procedure will show better blood pressure data during follow up, since the completeness has been assessed in contrast to the RNS-checked RDN procedure.

Study design: Investigator initiated, single centre, prospective, feasibility study

Study population: 40 patients (18 - 80 yr old)

* 20 patients treated with RNS-checked RDN
* 20 patients treated with RNS-guided RDN

Intervention:

Two different techniques will be used in this trial:

1. RNS-checked RDN
2. RNS-guided RDN

Main study endpoints:

Main study parameter will be the arterial blood pressure response to RNS prior to RDN and absence of blood pressure rise in response to pacing in the renal artery after RDN.

Secondary study endpoints:

Blood pressure at 3, 6, 12 months after the intervention, and change in blood pressure compared to measurement before the intervention.

ELIGIBILITY:
Inclusion Criteria:

* The patient is willing and able to comply with the protocol and has provided written informed consent.
* Age 18-80 years
* The patient has hypertension and is accepted for renal denervation or combined pulmonary bein isolation and renal denervation
* Glomerular filtration rate >45 mL/min
* No history of renal artery stenosis

Exclusion Criteria:

* Type 1 diabetes mellitus
* Contraindication to chronic anticoagulation therapy or heparin.
* Chronic oxygen use
* Primary pulmonary hypertension
* Woman currently pregnant or breastfeeding or not using reliable contraceptive measures during fertile age.
* Known secondary cause of hypertension
* Mental or physical inability to participate in the study.
* Renal artery stenosis >50% of the arterial lumen, or renal artery lumen ≤3 mm.
* Dual or triple ipsilateral renal artery ostia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2014-03-14 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2019-07-04 (Actual)

PRIMARY OUTCOMES:
arterial blood pressure response | during procedure
  Main study parameter will be the arterial blood pressure response to RNS prior to renal denervation and absence of blood pressure rise in response to pacing in the renal artery after RDN.

SECONDARY OUTCOMES:
blood pressure at 3 months | 3 months after the intervention
  Blood pressure at 3 months after the intervention
blood pressure at 6 months | 6 months after the intervention
  Blood pressure at 6 months after the intervention
blood pressure at 12 months | 12 months after the intervention
  Blood pressure at 12 months after the intervention
change in blood pressure compared to measurement before the intervention | intervention - up to 12 months after the intervention
  change in blood pressure compared to measurement before the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- A. Elvan, Zwolle, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hoogerwaard AF, Adiyaman A, de Jong MR, Smit JJ, Heeg JE, van Hasselt BAAM, Elvan A. Renal nerve stimulation: complete versus incomplete renal sympathetic denervation. Blood Press. 2021 Dec;30(6):376-385. doi: 10.1080/08037051.2021.1982376. Epub 2021 Oct 14. PMID 34647513